CLINICAL TRIAL: NCT03897413
Title: An Open-label, Randomized, Three-period, Crossover Study to Assess the Effect of Food and Calcium on S-888711 0.25-mg Tablet Pharmacokinetics in Healthy, Adult Volunteer Subjects Following a Single 0.75-mg Oral Dose of S-888711
Brief Title: Effect of Food and Calcium on Pharmacokinetics of a Single Dose of S-888711 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0924M0618
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence 1 (Experimental): Participants received a single oral dose of 0.75 mg S-888711 in the fasted state in treatment period 1, a single oral dose of 0.75 mg S-888711 in the fed state in period 2, and a single oral dose of 0.75 mg S-888711 in the fasted state with 4000 mg of calcium carbonate in period 3. Each period consisted of 6 days, separated by a 5-day washout period.
  Interventions: Drug: S-888711; Dietary Supplement: Calcium Antacid
- Sequence 2 (Experimental): Participants received a single oral dose of 0.75 mg S-888711 in the fed state in treatment period 1, a single oral dose of 0.75 mg S-888711 in the fasted state with 4000 mg of calcium carbonate in period 2, and a single oral dose of 0.75 mg S-888711 in the fasted state in period 3. Each period consisted of 6 days, separated by a 5-day washout period.
  Interventions: Drug: S-888711; Dietary Supplement: Calcium Antacid
- Sequence 3 (Experimental): Participants received a single oral dose of 0.75 mg S-888711 in the fasted state with 4000 mg of calcium carbonate in treatment period 1, a single oral dose of 0.75 mg S-888711 in the fasted state in period 2, and a single oral dose of 0.75 mg S-888711 in the fed state in period 3. Each period consisted of 6 days, separated by a 5-day washout period.
  Interventions: Drug: S-888711; Dietary Supplement: Calcium Antacid

INTERVENTIONS:
Drug: S-888711 — Administered orally as three 0.25 mg tablets
Dietary Supplement: Calcium Antacid — Calcium carbonate 4000 mg chewable tablets

SUMMARY:
The primary objectives of this study were:

* To assess the effect of a high-fat diet on the pharmacokinetics (PK) of a 0.75 mg single dose of S-888711 orally administered as 0.25 mg tablets in healthy volunteer adults
* To assess the effect of a calcium supplement on the PK of a 0.75 mg single dose of S-888711 orally administered as 0.25 mg tablets in healthy volunteer adults

ELIGIBILITY:
Inclusion Criteria:

1. A signed and dated written informed consent obtained prior to Screening.
2. Males and females ≥ 18 and ≤ 70 years of age, inclusive (at the time of informed consent).
3. Judged healthy at screening examination by the investigator.
4. Body mass index (BMI) of ≥ 19 to ≤ 29.9 kg/m².
5. All subjects must have agreed to use 2 forms of barrier contraception if engaging in sexual intercourse for at least 7 days prior to the first dose of study drug and continuing throughout the study, excluding subjects who had been surgically sterilized or females who had been postmenopausal (confirmed by follicle stimulating hormone test levels) for at least 1 year.
6. All female subjects must have had a negative urine pregnancy test.
7. Platelet count of 100,000 to 325,000/μL.
8. Willing to submit to blood sampling for the planned PK analysis.

Exclusion Criteria:

1. The use of prescription or non-prescription drugs, including herbal medicine or dietary supplements, within 14 days prior to dosing, with the exception of up to 3 doses of acetaminophen ≤ 1 gram each permitted from 14 days prior to the first study drug dose through 72 hours prior to the first study drug dose.
2. A history of regular use of tobacco- or nicotine-containing products within 6 months prior to Screening as confirmed by a urine cotinine test.
3. A history of use of inhibitors or inducers of cytochrome P450 (CYP) 3A4 within 14 days prior to Screening.
4. A history of use of platelet aggregation inhibitors, coronary artery vasodilators, calcium antagonists, beta blockers, diuretics, psychotropic drugs, prostaglandins, antibiotics, anticoagulants, and anticlotting or antiplatelet drugs (including aspirin and non-steroidal anti-inflammatory drugs) within 4 weeks prior to Screening.
5. History of use of thrombocytopenia-inducing drugs (eg, quinidine, trimethoprim sulfamethoxazole, etc.) within 4 weeks prior to Screening.
6. Family history of a hematologic disorder.
7. Hemorrhagic tendency.
8. A history of cardiac episode(s) or abnormal finding on electrocardiogram (ECG) and judged as ineligible by the investigator.
9. Chronic disease requiring medication and/or other treatment such as dietary restriction and physical therapy.
10. A history of anaphylaxis or significant side effect induced by a drug.
11. A history of allergic symptoms including food allergy, but excluding inactive pollen allergy.
12. A history of abuse of alcohol and/or drugs.
13. Positive urine screen for drug abuse.
14. A history of gastrointestinal surgery making subject ineligible as judged by the investigator.
15. Judged ineligible for this study by the investigator due to a history or clinical manifestations of significant metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, or urological disease or other clinically important disorder.
16. Positive laboratory results for hepatitis A IgM antibody, hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus at Screening.
17. Donation of >400 mL of blood within 12 weeks or >200 mL of blood within 4 weeks prior to Screening.
18. Prior administration of S-888711.
19. Use of other investigational products within 30 days or 6 half-lives (whichever was longer) prior to the first dose of study medication.
20. Judged ineligible for this study by the investigator for any other reason.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-11-06 (Actual); Primary Completion 2009-12-23 (Actual); Study Completion 2009-12-23 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration of S-888711 | Predose and 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours after dosing
Time to Maximum Observed Plasma Concentration of S-888711 | Predose and 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours after dosing
Area Under the Concentration-time Curve from Time Zero to the Time Point of the Last Quantifiable Concentration of S-888711 | Predose and 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours after dosing
Area Under the Concentration-time Curve from Time Zero to Infinity of S-888711 | Predose and 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours after dosing
Terminal Elimination Half-life of S-888711 | Predose and 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours after dosing
Apparent Total Clearance of S-888711 | Predose and 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours after dosing

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events | up to 40 days

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (1):
- Healthcare Discoveries, LLC, San Antonio, Texas, United States

REFERENCES:
- [Derived] Katsube T, Wajima T, Fukuhara T, Kano T. Effects of Food and Calcium Carbonate on the Pharmacokinetics of Lusutrombopag, a Novel Thrombopoietin Receptor Agonist. Clin Ther. 2019 Sep;41(9):1747-1754.e2. doi: 10.1016/j.clinthera.2019.06.004. Epub 2019 Jul 11. PMID 31303281